CLINICAL TRIAL: NCT00910546
Title: Image Guided and Breathing Adapted Radiotherapy of Early Stage Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gitte Fredberg Persson (Other)
Responsible Party: Sponsor-Investigator, Gitte Fredberg Persson, MD PhD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HPCRT002; H-B-2007-016 (Other: regional videnskabsetisk komite)
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Stereotactic radiotherapy; Image guidance; breathing adaption; tumor motion; implanted marker
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implantation of gold marker (Experimental): CT guided implantation of gold marker into early stage lung tumors. Extra 4DCT scans and fluoroscopies during planning and the 3 fraction radiotherapy course.
  Interventions: Device: visicoil gold marker 0.7 x 20 mm

INTERVENTIONS:
Device: visicoil gold marker 0.7 x 20 mm — CT - guided implantation into lung tumors
  Other Names: Gold Ancor

SUMMARY:
The purpose of this study is to quantify the variation in tumour middle position during a course of stereotactic body radiotherapy (SBRT), and thereby be able to design radiotherapy margins that takes into account the full motion span throughout an entire course of SBRT.

DETAILED DESCRIPTION:
Lung tumours move with respiration. This must be considered when designing margins for radiotherapy. This movement can be quantified by fluoroscopy or 4DCT. It is possible to identify a tumour middle position for planning. This middle position will vary from day to day and the extent of this variation is not fully known. The aim of this study is to quantify the variation in tumour middle position during a course of stereotactic body radiotherapy (SBRT), and thereby be able to design margins for patients that take into account the full motion span throughout an entire course of SBRT Patients: 15 consecutive patients with inoperable low stage lung cancer or solitary metastases to the lung (1-2) referred for SBRT - 45 Gy/3 fractions.

Methods: A gold coil will be implanted into the lung tumour one week before the planning. At planning and all treatment days supplementary 4DCT of thorax and two orthogonal fluoroscopy sessions will be performed. Tumour motion in the superior-inferior, medio-lateral and cranio-caudal direction will be measured and variation in amplitude and baseline for the tumour motion will be reported.

Perspective: By examining the variation in tumour movement it will be possible design margins for SBRT, accounting for the full tumour motion span and minimizing the risk of geographical miss and thereby optimizing the chance for local tumour control.

ELIGIBILITY:
Inclusion Criteria:

* tumor > 6 cm
* no more than 2 tumours
* histological proven non small celled lung cancer
* signed Informed Consent

Exclusion Criteria:

* Serious bleeding disorder
* Performance status 3-4
* Tumour close to large vessels (judged by interventional radiologist)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
motion of lung tumours | 3 weeks
  measured on 4DCT

SECONDARY OUTCOMES:
toxicity of implanting gold coils into lung tumours | 1 year
  complication rate

CONTACTS AND LOCATIONS:
Overall Officials: Gitte F Persson, MD, Principal Investigator — Rigshospitalet, Denmark; Ditte E Nygaard, MSc, Study Chair — Rigshospitalet, Denmark; Stine S Korreman, MSc PhD, Study Chair — Rigshospitalet, Denmark; Lena Specht, MD DMSc, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Department of Radiation Oncology, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No